CLINICAL TRIAL: NCT05924360
Title: The Impact of Mulligan and Maitland Techniques on Pain, Functionality, Proprioception, and Quality of Life in Individuals With Rotator Cuff Lesions
Brief Title: Impact of Mulligan and Maitland Techniques on Rotator Cuff Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, burak menek, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E-10840098-772.02-1672
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Rotator Cuff Tears
Keywords: Rotator cuff; Mulligan mobilization; Maitland mobilization; Exercise
MeSH Terms: conditions — Rotator Cuff Injuries; Motor Activity | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Other): The individuals in this group will undergo a conventional exercise program.
  Interventions: Other: conventional exercise program; Device: TENS
- Mulligan Group (Experimental): In addition to the conventional treatment program, individuals in this group will receive the mobilization with movement technique in the directions of flexion, abduction, and external rotation, twice a week.
  Interventions: Other: conventional exercise program; Other: Mulligan application
- Maitland Group (Experimental): In addition to the conventional treatment program, The Maitland application will be administered in the anterior-posterior, posterior-anterior, and caudal directions. The Maitland application will be delivered at grades 2-3. Patients in this group will receive the application in five sets of 30 seconds, twice a week.
  Interventions: Other: conventional exercise program; Other: Maitland application

INTERVENTIONS:
Other: conventional exercise program — The conventional treatment program will be applied to all participants included in the study, consisting of wand, codman, active and passive stretching exercises. This program will be administered to all patients five days a week. Wand exercises will be applied in the directions of flexion, abduction, extension, internal and external rotation, and will consist of 10 repetitions. Codman exercises will be applied in the directions of flexion, abduction, and circular, and will also consist of 10 repetitions. Active and passive stretching exercises will be applied in the directions of flexion, abduction, and external rotation, and will consist of 10 repetitions.
Other: Mulligan application — The mobilization with movement technique, a part of Mulligan applications, will be performed twice a week in the directions of flexion, abduction, and external rotation.
  Arms: Mulligan Group
Other: Maitland application — Maitland Group: The Maitland application will be applied in the anterior-posterior, posterior-anterior, and caudal directions. The Maitland application will be administered at grades 2-3. Patients in this group will receive the application in five sets of 30 seconds, twice a week.
  Arms: Maitland Group
Device: TENS — TENS application will be administered for 20 minutes at 100Hz
  Arms: Control Group

SUMMARY:
The shoulder joint in the human body has a broader range of motion and opening compared to other joints, resulting in a multitude of potential problems. The rotator cuff lesion is one such issue. The rotator cuff is found in the subacromial space of the shoulder and results from the compression of the subacromial bursa and the long head of the M.biceps muscle between the humerus and the coracoacromial arch.

Upon reviewing the literature, therapeutic exercise and electrotherapy modalities are the most preferred and studied areas. Alongside these, we also observe the usage of Mulligan and Maitland techniques for the treatment of rotator cuff lesions.

The Mulligan technique was developed by Brian Mulligan in 1980, who lent his name to it. Also known as mobilization with movement, this technique is often applied to the body's distal joints. The Maitland mobilization technique is used to treat the relevant joint with specific methods, particularly focusing on pain and stiffness in the joint. The technique's application is graded from 1 to 4. Grade 1 is a small oscillation created without loading throughout the joint movement. Grade 2 is performed with a slightly more oscillation from the beginning of the movement. Grades 1 and 2 aim to restrict the pain stimulus going to the central nervous system by stimulating the mechanoreceptor in the joint, thereby reducing the sensation of pain.

Grade 3 is applied at a larger amplitude until a limitation is felt from the middle of the joint movement. Lastly, grade 4 is applied to the limited small amplitude until tissue resistance is felt. Grades 3 and 4 are used to alleviate joint stiffness by applying shorter oscillation stimuli to a shorter tissue. The results of the use of Mulligan and Maitland techniques have been demonstrated in different studies in the literature. However, as far as we know, no study in the literature compares these two techniques in individuals with rotator cuff lesions. Based on this gap in the literature, the purpose of this study is to investigate the effects of the Mulligan technique and the Maitland method on pain, range of joint motion, functionality, joint position sense, and quality of life in individuals with a rotator cuff problem.

DETAILED DESCRIPTION:
The aim of this study is to examine the effectiveness of the Mulligan and Maitland techniques on pain, range of joint motion, functionality, joint position sense, and quality of life in individuals diagnosed with rotator cuff lesions. Individuals diagnosed with a rotator cuff lesion and admitted to Medipol University Hospital will be included in the study. Participants will be randomly divided into three groups. A conventional treatment program will be applied to individuals in all three groups five days a week for three weeks. The first group will only receive conventional treatment. The second group will receive conventional treatment plus the Mulligan technique. The third group will receive conventional treatment plus the Maitland technique. The conventional treatment program will be applied to all participants included in the study, consisting of wand, codman, active and passive stretching exercises, and TENS. This program will be administered to all patients five days a week. Wand exercises will be applied in the directions of flexion, abduction, extension, internal and external rotation, and will consist of 10 repetitions. Codman exercises will be applied in the directions of flexion, abduction, and circular, and will also consist of 10 repetitions. Active and passive stretching exercises will be applied in the directions of flexion, abduction, and external rotation, and will consist of 10 repetitions. TENS application will be administered for 20 minutes at 100Hz. All these exercises will be applied to the control, Mulligan, and Maitland groups.

Mulligan Group: The mobilization with movement technique, a part of Mulligan applications, will be performed twice a week in the directions of flexion, abduction, and external rotation.

Maitland Group: The Maitland application will be applied in the anterior-posterior, posterior-anterior, and caudal directions. The Maitland application will be administered at grades 2-3. Patients in this group will receive the application in five sets of 30 seconds, twice a week.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 30 and 70
* Not having undergone any previous shoulder surgery
* Being diagnosed with a rotator cuff lesion
* Not having any orthopedic or cardiac problems that could interfere with the study or evaluation

Exclusion Criteria:

* Having a pathology affecting the shoulder region
* Having undergone any shoulder surgery
* Individuals who are not cooperative or have mental problems
* Individuals with neurological, cardiac, and vascular problems
* Individuals who have participated in any physiotherapy program targeting the shoulder in the past 3 months

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-26 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 5 minutes
  Visual Analog Scale (VAS) The Visual Analog Scale is a commonly preferred evaluation method in clinical practice and literature studies for measuring pain intensity. Patients' pain levels are determined by numbering the range from 0 to 10. A score of 0 indicates no pain, while 10 represents the most intense pain felt.
Range of Motion | 10 minutes
  Range of Joint Motion Evaluating the range of joint motion (ROM) is an objective method frequently used in both clinical settings and academic studies. The universal goniometer, used for assessing ROM, is the most preferred tool. In addition to determining the limit of joint movement, it is also used to provide clinicians with data on the effectiveness of the treatment.
Joint Postion Sense | 5 minutes
  The joint position sense measurements of the individuals participating in the study will be evaluated using a goniometer. Participants will be asked to raise their shoulder to a certain degree, and then return it to the same angle with their eyes closed. The angular value formed when the eyes are closed and open will be recorded, and the difference between the shoulder angles will be calculated. The joint position sense will be applied at 30 and 60 degrees of flexion and abduction movements.

SECONDARY OUTCOMES:
Disabilities of the Arm, Shoulder, and Hand Questionnaire | 10 minutes
  The DASH (Disabilities of the Arm, Shoulder and Hand) outcome measure is a result of collaborative efforts by the American Academy of Orthopedic Surgeons and other organizations, designed to evaluate physical limitations and function in upper extremity lesions. The DASH questionnaire consists of three subsections. The first part includes 30 questions; 21 questions assess the difficulties encountered in the patient's daily life functions, 5 questions evaluate symptoms, and the remaining 4 questions assess social life, work, sleep, and self-confidence of the individual. The four-question section, also known as the Work Module (DASH-WM), which can be answered optionally, measures the difficulties the individual encounters in their work life.
Rotator cuff quality of life | 10 minutes
  The quality of life scale developed by Hollinshead et al. is a measure that allows the participant to evaluate their own quality of life. Comprising a total of 34 questions, the scale consists of five sections evaluating disease symptoms and physical complaints (16 questions), work/occupation activities (4 questions), leisure activities (4 questions), lifestyle (5 questions), and social and emotional aspects (5 questions). Each question is answered with a 100 mm visual analog scale: "0" indicates the lowest and "100" the highest score. The total score is then represented as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Burak Menek, PhD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No